CLINICAL TRIAL: NCT02395224
Title: A Longitudinal Study of Colorectal Cancer Patients With Metastatic Disease in Middle-Norway
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Midt-Norge (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/1361
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Neoplasms, Colorectal; Neoplasm Metastasis
Keywords: Follow-up studies; Prognosis; Palliative care; Chemotherapy, adjuvant; Cost-benefit analysis; Population; Antineoplastic agents/Adverse effects; Terminal care; Medical futility; Survival rate; Norway
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: cancer treatment and follow-up according to current regional and national guidelines

SUMMARY:
The main objective is to provide original research results that may change clinical practice related to metastatic colorectal cancer. The study will evaluate treatment and patient care at different stages of the disease trajectory and the use of health care for this large group of patients. It will be possible to compare the effectiveness of chemotherapy, radiotherapy and symptomatic treatment given to "real life" patients with the efficacy reported in randomised clinical trials. By using longitudinal information on imaging, biomarkers, clinical staging and place of care it will be possible to improve patient classification at various stages of the disease. Based on this, a more appropriate, individualized treatment for colorectal cancer may be recommended during the phases of the disease trajectory. Participation in this project will not influence the treatment for colorectal cancer. All patients will be treated and followed-up according to current regional and national guidelines.

DETAILED DESCRIPTION:
The available evidence-based knowledge of patient management is translated into regularly updated clinical guidelines for diagnosis, staging and treatment. The guidelines represent the basis for oncology care in Norway, and health care providers are expected to follow these guidelines. Current guidelines are derived from studies where patients are highly selected and not representative for the whole cohort of patients with metastatic disease. One can speculate if the results of trials conducted in regional centers can be generalized to whole populations in a region. In this respect it will be valuable to study advanced colorectal cancer in the whole population of Middle-Norway, with both one regional center and all other hospitals in the area. More knowledge is needed for the optimal selection of treatment for individual patients. In relation to symptom relief, physical and psychological functioning and overall quality of life, there is clearly a lack of high quality research.

A longitudinal follow-up of a large number of metastatic colorectal cancer patients with regular assessments has not been previously launched. The existing infrastructure in Norway makes the study feasible and will provide high internal and external validity related to clinical outcomes. The study will constitute a unique platform for comprehensive research aimed at this patient group. It also provides a concept that can be transferred to other major diseases, and it can be extended to other health regions of Norway.

ELIGIBILITY:
Inclusion Criteria:

* Colon or rectal cancer with synchronous metastases.
* Colon or rectal cancer with metastatic relapse after curative primary treatment (for localized disease or maximum one operation for distant metastases)
* Localized colon or rectal cancer that due to tumor or patient related factors are not treated with a curative intent
* Written informed consent. In patients not able to consent due to cognitive impairment consent can be by proxy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosis of metastatic colorectal cancer treated with a curative or non-curative intention, or local disease not treated with a curative intention.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
survival | 3 years or until death
  Cancer-specific and overall survival according to treatment, age, sex, biological markers

SECONDARY OUTCOMES:
Nutritional status | 3 years or until death
  reported on PG-SGA, patient version
Patient expectations | 3 years or until death
  patient expectations about effects of chemotherapy and satisfaction with treatment
WHO performance status | 3 years or until death
Toxicity of therapy | 3 years or until death
  Number of dose reductions and treatment delays
Toxicity of therapy | 3 years or until death
  Common Terminology Criteria for Adverse Events (CTCAE) v4.0; grade 3-4 for the following items: Hematology, infectious, gastrointestinal, neurological and thromboembolism
Health related quality of life | 3 years or until death
  reported on EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD PhD, Study Director — Norwegian University of Science and Technology
Locations (7):
- Norway (7):
  - Ålesund Hospital, Ålesund
  - Kristiansund Hospital, Kristiansund
  - Levanger Hospital, Levanger
  - Molde hospital, Molde
  - Namsos Hospital, Namsos
  - St Olavs Hospital, Trondheim
  - Volda Hospital HF, Volda

REFERENCES:
- [Derived] Hatlevoll I, Kristensen AK, Solheim TS, Elvebakken H, Salvesen O, Oldervoll LM, Wibe A, Hofsli E. Do older patients with colorectal cancer experience more deterioration in health-related quality of life than younger patients during the first year of palliative chemotherapy? A prospective real-world observational study. J Geriatr Oncol. 2024 Apr;15(3):101715. doi: 10.1016/j.jgo.2024.101715. Epub 2024 Feb 15. PMID 38359528